## Youth Mayo Clinic Anxiety Coach Pilot Study

13-000288 - PILOT

NCT02205177

Date: July 1, 2019

The data were primarily analyzed descriptively. To demonstrate the potential of *Anxiety Coach* to monitor fidelity data on exposure use by session were examined by therapist. Similarly, to demonstrate the potential of *Anxiety Coach* to monitor patient engagement data on completed exposures were examined by patient and condition. To address technological issues that contributed to exposures being inaccurately recorded: a) those with zero seconds duration were removed (e.g., recording an exposure only to mark an item as mastered); b) those with an anxiety rating of zero at the beginning, all of which were five seconds in duration or less, were removed; c) exposures of less than an minute in duration that included an initial anxiety rating greater than zero were counted as exposures, but the duration was not entered in the average duration (e.g., recording previously completed exposures); d) exposures with durations of multiple hours were included in the exposure count, but not entered in the average duration. (e.g., suggesting that the program was left running unattended during an exposure. Symptom measure at pre- and post-treatment are presented by patient and condition to provide a preliminary examination of outcomes.

Semi-structured Interviews were conducted with five families using purposive sampling approach in which parents and children most likely to have informative opinions (positive or negative) and able to communicate them were selected among all agreeing to participate in the interview (all families were invited). All interviews were conducted by two qualitative researchers (JCH and KVD) not involved in the development or delivery of the app. Interviews were recorded and transcribed verbatim. Interviews concluded when data saturation was reached, and data were independently analyzed and compared using methods of content analysis, organized by predominant themes.